CLINICAL TRIAL: NCT04340193
Title: A Randomized, Multi-center, Double-blinded, Placebo-controlled Phase 3 Study of Nivolumab and Ipilimumab, Nivolumab Monotherapy, or Placebo in Combination With Trans-arterial ChemoEmbolization (TACE) in Patients With Intermediate-stage Hepatocellular Carcinoma (HCC)
Brief Title: A Study of Nivolumab and Ipilimumab and Nivolumab Alone in Combination With Trans-arterial ChemoEmbolization (TACE) in Participants With Intermediate Stage Liver Cancer
Acronym: CheckMate 74W
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-74W
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Cancer, Hepatocellular
MeSH Terms: conditions — Liver Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab + Ipilimumab + TACE (Experimental): TACE (Trans-arterial ChemoEmbolization)
  Interventions: Drug: nivolumab; Drug: ipilimumab; Procedure: TACE
- Nivolumab + TACE (Experimental)
  Interventions: Drug: nivolumab; Procedure: TACE
- TACE (Active Comparator)
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Nivolumab + Ipilimumab + TACE; Nivolumab + TACE
Drug: ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Nivolumab + Ipilimumab + TACE
Procedure: TACE — TACE (Trans-arterial ChemoEmbolization)

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of nivolumab with and without ipilimumab in combination with Trans-arterial ChemoEmbolization (TACE) to TACE alone in participants with intermediate liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant has intermediate-stage hepatocellular carcinoma (HCC) whose tumor characteristics exceed the Beyond Milan and Up-to-7 (BMU7) criteria and is eligible for trans-arterial ChemoEmbolization (TACE)
* Participant has no extrahepatic spreading (EHS), no regional lymph node involvement, no main, left main, or right main portal vein thrombosis, and no macrovascular invasion (MVI)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Prior liver transplant or participants who are on the waiting list for liver transplantation
* Active, known, or suspected autoimmune disease

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (105):
- United States (5):
  - Local Institution - 0189, Coronado, California
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution - 0005, Louisville, Kentucky
  - Local Institution - 0059, Louisville, Kentucky
  - Local Institution - 0109, Dallas, Texas
- Australia (5):
  - Local Institution, Wollongong, New South Wales
  - Local Institution - 0037, Birtinya, Queensland
  - Local Institution - 0010, Adelaide, South Australia
  - Local Institution - 0001, Melbourne, Victoria
  - Local Institution - 0139, Murdoch, Western Australia
- Austria (5):
  - Local Institution - 0026, Graz
  - Local Institution - 0013, Sankt Pölten
  - Local Institution, Vienna
  - Local Institution - 0078, West Springfield
  - Local Institution - 0048, Wiener Neustadt
- Belgium (4):
  - Local Institution - 0020, Brussels
  - Local Institution, Federal District
  - Local Institution - 0053, Ghent
  - Local Institution - 0050, Plainfield
- Local Institution - 0039, Québec, Quebec, Canada
- China (10):
  - Local Institution - 0184, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Tianjin, Hebei
  - Local Institution - 0196, Nanjing, Jiangsu
  - Local Institution - 0176, Nanchang, Jiangxi
  - Local Institution, Shenyang, Liaoning
  - Local Institution - 0209, Xi'an, Shan3xi
  - Local Institution - 0151, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Hangzhou, Zhejiang
- Czechia (2):
  - Local Institution - 0055, Olomouc
  - Local Institution, Prague
- France (12):
  - Local Institution - 0014, Lille, Mount
  - Local Institution - 0132, Caen
  - Local Institution - 0021, Clichy
  - Local Institution - 0064, Dijon
  - Local Institution - 0082, Englewood
  - Local Institution - 0052, La Tronche
  - Local Institution - 0061, Marseil
  - Local Institution - 0087, Nantes
  - Local Institution - 0012, Nice
  - Local Institution - 0093, Paris
  - Local Institution - 0046, Reims
  - Local Institution - 0094, Villejuif
- Germany (4):
  - Local Institution - 0035, Göttingen
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution - 0071, Leipzig
- Hong Kong (2):
  - Local Institution - 0004, Hong Kong
  - Local Institution - 0045, Hong Kong
- Italy (8):
  - Local Institution - 0015, Orbassano, TO
  - Local Institution, Messina
  - Local Institution - 0025, Milan
  - Local Institution, Monserrato
  - Local Institution, Parma
  - Local Institution, Roma
  - Local Institution - 0076, Siena
  - Local Institution - 0070, Vicenza
- Japan (15):
  - Local Institution - 0108, Chiba, Chiba
  - Local Institution - 0122, Matsuyama, Ehime
  - Local Institution - 0148, Sapporo, Hokkaido
  - Local Institution - 0118, Kanazawa, Ishikawa-ken
  - Local Institution - 0120, Yokohama, Kanagawa
  - Local Institution - 0113, Yokohama, Kanagawa
  - Local Institution - 0115, Kyoto, Kyoto
  - Local Institution - 0127, Abeno-ku, Osaka
  - Local Institution - 0125, Izunokuni-Shi, Shizuoka
  - Local Institution - 0116, Minato-ku, Tokyo
  - Local Institution - 0128, Minato-ku, Tokyo
  - Local Institution - 0121, Musashino-shi, Tokyo
  - Local Institution - 0119, Hiroshima
  - Local Institution - 0117, Osaka
  - Local Institution - 0123, Saitama
- Local Institution, Warsaw, Poland
- Local Institution - 0049, San Juan, Puerto Rico
- Russia (3):
  - Local Institution - 0016, Barnaul
  - Local Institution - 0077, Saint Petersburg
  - Local Institution - 0009, Saint Petersburg
- Singapore (3):
  - Local Institution - 0027, Singapore
  - Local Institution - 0089, Singapore
  - Local Institution - 0011, Singapore
- South Korea (8):
  - Local Institution - 0114, Busan
  - Local Institution - 0135, Daegu
  - Local Institution - 0047, Gyeongsangnam-do
  - Local Institution - 0097, Hwasun-Gun
  - Local Institution - 0161, Seoul
  - Local Institution - 0186, Seoul
  - Local Institution - 0160, Seoul
  - Local Institution - 0164, Seoul
- Spain (9):
  - Local Institution - 0023, Alicante
  - Local Institution - 0092, Córdoba
  - Local Institution - 0101, Madrid
  - Local Institution - 0183, Madrid
  - Local Institution - 0084, Madrid
  - Local Institution - 0018, Madrid
  - Local Institution - 0099, Pamplona
  - Local Institution - 0131, Sabadell
  - Local Institution - 0102, Santiago de Compostela
- Taiwan (7):
  - Local Institution - 0136, Buzi
  - Local Institution - 0141, Kaohsiung City
  - Local Institution - 0030, Taichung
  - Local Institution - 0057, Taichung
  - Local Institution - 0029, Tainan
  - Local Institution - 0002, Taipei
  - Local Institution - 0044, Tapei

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT04340193.html

RESULTS

PARTICIPANT FLOW:
Groups:
- NIVO+IPI+TACE: Participants with intermediate-stage hepatocellular carcinoma (HCC) received Nivolumab (NIVO) 240 milligram (mg) every 2 weeks (Q2W) and ipilimumab (IPI) 1 milligram per kilogram (mg/kg) every 6 weeks (Q6W) as an approximately 30-minute infusion. Participants received first Trans-arterial ChemoEmbolization (TACE) in 7 days after randomization and then TACE as needed, until participant was no longer eligible for further TACE, unacceptable toxicity, withdrawal of consent, or the study ends, whichever occurs first.
- NIVO+TACE: Participants with intermediate-stage hepatocellular carcinoma (HCC) received Nivolumab 240 milligram (mg) every 2 weeks (Q2W) as an approximately 30-minute infusion. Participants received first Trans-arterial ChemoEmbolization (TACE) in 7 days after randomization and then TACE as needed, until participant was no longer eligible for further TACE, unacceptable toxicity, withdrawal of consent, or the study ends, whichever occurs first. Per Protocol Amendment 01, participants did not receive placebo infusions following unblinding.
- TACE: Participants received first Trans-arterial ChemoEmbolization (TACE) in 7 days after randomization and then TACE as needed, until participant was no longer eligible for further TACE, unacceptable toxicity, withdrawal of consent, or the study ends, whichever occurs first. Per Protocol Amendment 01, participants did not receive placebo infusions following unblinding.
Period: Overall Study
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Started | 9 | 9 | 8
Completed | 6 | 4 | 4
Not Completed | 3 | 5 | 4
Not completed — Other reason | 0 | 0 | 1
Not completed — Disease recurrence | 0 | 1 | 0
Not completed — Study drug toxicity | 1 | 0 | 0
Not completed — Disease progression | 1 | 2 | 3
Not completed — Administrative reasons by sponsor | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE | Total
Number analyzed (Participants) | 9 | 9 | 8 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.3 (10.28) | 62.7 (11.19) | 70.3 (8.89) | 68.3 (10.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 7 | 8 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 4 | 4 | 8
  Unknown or Not Reported | 9 | 4 | 4 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 3 | 2 | 8
  Black or African American | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 3 | 4
  Chinese | 2 | 2 | 1 | 5
  Japanese | 2 | 1 | 2 | 5
  Not Reported | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants | 9 | 9 | 8

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose that results in death, Is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe) or requires inpatient hospitalization or causes prolongation of existing hospitalization, or results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect or is an important medical event.
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants | 7 | 6 | 2

3. Primary Outcome: Number of Participants Who Died
Description: Number of participants who died due to any cause are summarized.
Time Frame: From first dose and 100 days after last dose of study therapy (up to approximately 27 months)
Population: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants | 2 | 2 | 0

4. Primary Outcome: Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Description: as for outcome 1
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants | 3 | 1 | 1

5. Primary Outcome: Number of Participants With Worst Grade (Grade 3/4) Laboratory Results
Description: Laboratory results were graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 (Grade 3 =Severe, Grade 4 = Life-threatening). Highest grade measured for hemoglobin and albumin was Grade 3.
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants
  Hemoglobin (Grade 3) | 1 | 0 | 2
  Platelet count (Grade 3) | 2 | 0 | 0
  Platelet Count (Grade 4) | 0 | 0 | 0
  Leukocytes (Grade 3) | 1 | 0 | 0
  Leukocytes (Grade 4) | 0 | 0 | 0
  Lymphocytes (Grade 3) | 2 | 2 | 3
  Lymphocytes (Grade 4) | 1 | 0 | 0
  Aspartate Aminotransferase (Grade 3) | 2 | 0 | 0
  Aspartate Aminotransferase (Grade 4) | 1 | 0 | 0
  Alanine Aminotransferase (Grade 3) | 1 | 1 | 0
  Alanine Aminotransferase (Grade 4) | 1 | 0 | 0
  Bilirubin, Total (Grade 3) | 0 | 0 | 0
  Bilirubin, TOTAL (Grade 4) | 1 | 0 | 0
  Creatinine, (Grade 3) | 0 | 1 | 0
  Creatinine (Grade 4) | 0 | 0 | 0
  Potassium, (Grade 3) | 1 | 1 | 0
  Potassium (Grade 4) | 0 | 0 | 0
  Amylase (Grade 3) | 2 | 0 | 0
  Amylase (Grade 4) | 0 | 0 | 0
  Lipase (Grade 3) | 4 | 0 | 1
  Lipase (Grade 4) | 0 | 0 | 0
  Albumin, (Grade 3) | 1 | 0 | 0
  Absolute Neutrophil Count (Grade 3) | 0 | 0 | 0
  Absolute Neutrophil Count (Grade 4) | 0 | 0 | 0
  Alkaline Phosphatase (Grade 3) | 0 | 0 | 0
  Alkaline Phosphatase (Grade 4) | 0 | 0 | 0
  Sodium (Grade 3) | 0 | 0 | 0
  Sodium (Grade 4) | 0 | 0 | 0
  Calcium, Total (Grade 3) | 0 | 0 | 0
  Calcium, Total (Grade 4) | 0 | 0 | 0
  Magnesium (Grade 3) | 0 | 0 | 0
  Magnesium (Grade 4) | 0 | 0 | 0
  Glucose (Grade 3) | 0 | 0 | 0
  Glucose (Grade 4) | 0 | 0 | 0
  Hypernatremia (Grade 3) | 0 | 0 | 0
  Hypernatremia (Grade 4) | 0 | 0 | 0
  Hyponatremia (Grade 3) | 0 | 0 | 0
  Hyponatremia (Grade 4) | 0 | 0 | 0
  Hyperkalemia (Grade 3) | 0 | 0 | 0
  Hyperkalemia (Grade 4) | 0 | 0 | 0
  Hypokalemia (Grade 3) | 1 | 1 | 0
  Hypokalemia (Grade 4) | 0 | 0 | 0
  Hypercalcemia (Grade 3) | 0 | 0 | 0
  Hypercalcemia (Grade 4) | 0 | 0 | 0
  Hypermagnesemia (Grade 3) | 0 | 0 | 0
  Hypermagnesemia (Grade 4) | 0 | 0 | 0
  Hypomagnesemia (Grade 3) | 0 | 0 | 0
  Hypomagnesemia (Grade 4) | 0 | 0 | 0
  Hypoglycemia (Grade 3) | 0 | 0 | 0
  Hypoglycemia (Grade 4) | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Blood samples were collected for specific thyroid test.
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants with at least one on-treatment thyroid stimulating hormone (TSH) measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants
  TSH > ULN (Upper Limit of Normal) | 5 | 5 | 5
  TSH > ULN with TSH <= ULN at baseline | 5 | 4 | 3
  TSH > ULN with at least one FT3/FT4 test value < LLN (Lower Limit of Normal) | 3 | 1 | 3
  TSH > ULN with all other FT3/FT4 test values >= LLN | 5 | 4 | 4
  TSH > ULN with FT3/FT4 test missing | 0 | 2 | 1
  TSH < LLN | 3 | 1 | 0
  TSH < LLN with TSH >= LLN at baseline | 3 | 1 | 0
  TSH < LLN with at least one FT3/FT4 test value > ULN | 2 | 0 | 0
  With all other FT3/FT4 test values <= ULN | 3 | 0 | 0
  With FT3/FT4 test missing | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities in Specific Liver Tests
Description: Blood samples were collected for specific liver tests.
Time Frame: From first dose and 30 days after last dose of study therapy (up to approximately 25 months)
Population: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
Number analyzed (Participants) | 9 | 9 | 8
Participants
  ALT or AST > 5 X Upper limit of Normal (ULN) | 3 | 2 | 0
  Alanine Transaminase (ALT) or AST > 10 X ULN | 2 | 1 | 0
  ALT or Aspartate Transaminase (AST) > 20 X ULN | 1 | 0 | 0
  Total Bilirubin > 2 X ULN | 3 | 2 | 1
  ALP (Alkaline Phosphatase) > 1.5 X ULN | 5 | 5 | 5
  Concurrent ALT OR AST Elevation > 3 X ULN with total Bilirubin > 2 X ULN within one day | 3 | 1 | 0
  Concurrent ALT or AST elevation > 3 X ULN with total Bilirubin > 2 X ULN within 30 days | 3 | 2 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from randomization until their study completion (up to approximately 38 months). Serious and non-serious adverse events were collected from first dose to 100 days after last dose of study therapy (up to approximately 27 months).
Description: All treated participants included all enrolled participants who received at least one dose of any study treatment.
Arm/Group | NIVO+IPI+TACE | NIVO+TACE | TACE
All-Cause Mortality (participants affected / at risk) | 2/9 | 2/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 7/9 | 6/9 | 2/8
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIVO+IPI+TACE (N=9) | NIVO+TACE (N=9) | TACE (N=8)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic infection (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0
Cell death (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 2 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NIVO+IPI+TACE (N=9) | NIVO+TACE (N=9) | TACE (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 4
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 2
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 2
Portal hypertensive gastropathy (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 2 | 2 | 1
Device related thrombosis (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 3
Pyrexia (General disorders) | 2 | 3 | 2
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Dermo-hypodermitis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 1
Genital herpes (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatobiliary procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post embolisation syndrome (Injury, poisoning and procedural complications) | 2 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0
Blood creatinine increased (Investigations) | 2 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Gastric pH decreased (Investigations) | 1 | 0 | 0
Inflammatory marker increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 4 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT04340193/Prot_SAP_000.pdf